CLINICAL TRIAL: NCT05091632
Title: Can You Hear Me? Assessment of Verbal Comprehension and Cognitive Processes in Patients in the Last Days of Life
Brief Title: Assessment of Verbal Comprehension and Cognitive Processes in Patients Admitted to the Palliative and Supportive Care Unit
Status: Suspended | Type: Observational
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1079; NCI-2021-08958 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1079 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-28; First posted 2021-10-25 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Observational (EEG, questionnaires): Patients undergo EEG over 30 minutes daily until death or discharge and complete questionnaires over 30 minutes daily until death or discharge to check level of consciousness, thought, and ability to communicate.
  Interventions: Procedure: Electroencephalography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Electroencephalography — Undergo EEG
  Other Names: EEG; electroencephalogram
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study investigates the use electroencephalography (EEG - a test that measures brain waves) to learn if patients who appear unresponsive (do not respond to noises, words, or touch) retain any consciousness. Families want to know if their loved ones who are unresponsive can still hear them or feel any discomfort. Information gained from this study may have important impact in how patients, caregivers, and doctors make decisions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the magnitude of electroencephalography (EEG) response to verbal stimuli among cancer patients in the last days in life admitted to a palliative and supportive care unit (PSCU).

II. To examine the feasibility of conducting EEG in cancer patients in the last days of life.

SECONDARY OBJECTIVES:

I. To compare the magnitude of EEG response between impending death cohort and control cohort.

II. To determine the association between the magnitude of EEG response and clinical assessments (e.g. JFK Coma Recovery Scale-Revised [CRS-R], Glasgow Coma Scale [GCS], Richmond Agitation Sedation Scale [RASS], Memorial Delirium Assessment Scale [MDAS]) in impending death cohort and control cohort separately.

III. To determine the magnitude of EEG response to pressure/noxious stimuli in impending death cohort and control cohort separately.

IV. To examine serial EEG changes in auditory cortex activation and cognitive processing in cancer patients over the last days of life.

OUTLINE:

Patients undergo EEG over 30 minutes daily until death or discharge and complete questionnaires over 30 minutes daily until death or discharge to check level of consciousness, thought, and ability to communicate.

ELIGIBILITY:
Inclusion Criteria:

1. [Both cohorts] Diagnosis of advanced cancer (defined as locally advanced, metastatic, recurrent, or incurable disease)
2. [Both cohorts] Admitted to the PSCU at MD Anderson Cancer Center or seen by the specialist palliative care inpatient consultation team (control cohort only)
3. [Impending death cohort] Clinician judgement of .3 days of survival or .1 late sign of impending death*
4. [Impending death cohort] Palliative Performance Scale score of 10-20%
5. [Control cohort] Able to communicate for the past 24 hours
6. [Control cohort] Clinician judgement of .1 month of survival
7. [Both cohorts] English-speaking

Exclusion Criteria:

1. [Both cohorts] Hearing impairment that significantly impacts daily communication with caregiver prior to entering impending death phase OR requiring hearing aid
2. [Impending death cohort] Mental status changes only related to medications as per clinician judgement
3. [Control cohort] Diagnosis of delirium (i.e. MDAS .13)
4. [Both cohorts] Pregnant women
5. [Both Cohorts] Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer admitted to the palliative and supportive care unit at M.D. Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Magnitude of electroencephalography (EEG) response to verbal stimuli among impending death cancer patients | Day 1 in palliative and supportive care unit
  The magnitudes of EEG responses in each task will be calculated as the difference between pre-stimulus and post-stimulus, separately. 95% confidence intervals will be estimated for each task.

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org